CLINICAL TRIAL: NCT05172635
Title: Primary Tumour Response to Induction Chemotherapy in Synchronously Metastasized Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Klinik Favoriten (Other)
Responsible Party: Principal Investigator, Thomas Gruenberger, Prim. Prof. Dr. med., Klinik Favoriten
Other Study IDs: 0001
Record Dates: First submitted 2021-11-28; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Gastrointestinal Neoplasm
Keywords: colorectal cancer; synchronous liver metastases; targeted therapy; tumour regression grading
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients, who received a VEGF antibody: We distinguished between patients who received a VEGF antibody therapy and patients who received a EGFR antibody therapy.
- Patients, who received a EGFR antibody: We distinguished between patients who received a VEGF antibody therapy and patients who received a EGFR antibody therapy.

SUMMARY:
We performed a retrospective data analysis of patients with synchronously metastasized colorectal cancer, comparing the histological response on the primary tumour to chemotherapy combined with either vascular endothelial growth factor (VEGF) or epidermal growth factor receptor (EGFR) inhibition.

DETAILED DESCRIPTION:
We performed a retrospective analysis regarding the response of the primary tumour and the liver metastases of patients with colorectal carcinoma to an induction chemotherapy with antibody therapy, either with a VEGF antibody, or with an EGFR antibody.

We investigated 100 Patients with synchronous metastatic colorectal carcinoma, who underwent hepatic resection in Clinic Landstraße or Clinic Favoriten between 2014 and 2021.

We investigated the tumour response of the primary tumour, using Rödel score, which is a tumour regression score.

We also investigated the tumour response of the liver metastases using Rubbia Brandt tumour regression score.

The pathological response was assessed postoperatively in the surgical specimen. In order to ensure a uniform assessment, the pathologists in our HPB center assessed the histological specimens from both treatment locations prior to this analyses.

The tumour response of the liver metastases was assessed twice: by radiological tumour assessment via computer tomography (CT) of the abdomen or magnetic resonance imaging (MRI) of the liver with RECIST criteria.

Postoperative complications less than 90 days after liver resection were assessed and described according to the classification system by Dindo et al.

Day of tumour recurrence and/or death was assessed.

We also investigated the difference of recurrence free Survival (RFS) and Overall surcical (OS) between the patients, who received EGFR and the patients, who received VEGF antibody treatment.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* synchronously hepatic metastasized patients with colorectal carcinoma
* indication of surgical treatment

Exclusion Criteria:

* younger than 18 years
* metachronously metastasized patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients had synchronously metastasized colorectal cancer and received surgical treatment because of their liver metastases in either Clinic Landstrasse or Clinic Favoriten (HPB center) in Vienna from June 2014 to February 2021..
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Pathological response of the primary tumour | Tumour regression was assessed in the surgical specimen 3 to 7 days after surgery.
  Investigation of the tumour response of the primary tumor (colorectal carcinoma) using the Rödel Score (tumour regression score)

SECONDARY OUTCOMES:
Pathological response of the liver metastases | Tumour regression was assessed in the surgical specimen 3 to 7 days after surgery. Radiological response was assessed in staging CT abdomen 2 to 4 weeks after induction chemotherapy.
  Investigation of the tumour response of the liver metastases using Rubbia Brand score (Tumour regression score) and using radiological assessment
Overall survival | median of 21 months (0 to 80)
  Difference of overall survival between patients, who received VEGF antibody treatment and patients, who received EGFR antibody treatment
Recurrece free survival | median of 21 months (0-80)
  Difference of recurrence free survival between patients, who received VEGF antibody treatment and patients, who received EGFR antibody treatment
90 day mortality | 90 days
  number of patients, who died less than 90 days after liver surgery

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gruenberger, Prof. Dr. med., Principal Investigator — Clinic Favoriten (HPB center)
Locations (1):
- Clinic Favoriten, Vienna, Vienna/Austria, Austria

IPD SHARING:
Plan to Share IPD: Undecided